CLINICAL TRIAL: NCT06784271
Title: Effect of Acute Phenylcapsaicin Intake on Trained Cross-Training Athletes: a Randomized, Placebo-Controlled Crossover Study
Brief Title: Effect of Acute Phenylcapsaicin Intake on Trained Cross-Training Athletes
Acronym: CROSSCAPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Universidad de La Laguna, San Cristóbal de La Laguna, Santa Cruz de Tenerife, Spain. (Unknown)
Responsible Party: Principal Investigator, Lucas Jurado-Fasoli, PhD, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CROSSCAPS
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Performance
Keywords: Phenylcapsaicin; performance; concurrent exercise; nutrition; recovery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phenylcapsaicin (Experimental): 2.5 mg of Phenylcapsaicin
  Interventions: Dietary Supplement: Phenylcapsaicin
- Placebo (Placebo Comparator): Preparation of colorants, sweeteners, aromas, and acidulants
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Phenylcapsaicin — 2.5mg of Phenylcapsaicin
  Arms: Phenylcapsaicin
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the effect of acute phenylcapsaicin intake during a cross-training session on perceived exertion, performance, and recovery in cross-training athletes.

DETAILED DESCRIPTION:
Capsaicin appears to enhance athletic performance by reducing perceived effort, increasing mechanical performance (e.g., total volume load), and decreasing muscle damage. Given the close relationship between the metabolic and physiological responses of cross-training and supplementation with Phenylcapsaicin (PC), it could be expected that consuming capsaicin during cross-training would have a favorable impact on perceived effort, recovery, and performance.

25 women and 24 men trained in CrossFit consumed either Phenylcapsaicin (PC) or a placebo during a CrossFit class, which consisted of a 16-minute weightlifting segment and a 15-minute WOD. Both the Rating of Perceived Exertion (RPE) and the Perceived Recovery Status scale (RPS) were administered at the beginning of the session and at the end of each segment of the CrossFit session. DOMS was assessed using a visual analog scale at 24 and 48 hours after the CrossFit session.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years.
* Body mass index: 18.5-30 kg/m2.
* Ability to understand the instructions, objectives, and study protocol.
* Minimum of 3 years of experience in crosstraining, with at least 6 hours of weekly training over the past 3 months.
* Resident on the island of Tenerife.

Exclusion Criteria:

* History of a significant adverse cardiovascular event, renal insufficiency, cirrhosis, eating disorder, weight control surgical intervention, or type 2 diabetes mellitus.
* Any chronic pathology in which the intake of nutritional supplements, especially pungent components, is not recommended.
* Any condition that, in the investigator's judgment, would impair the ability to participate in the study or represent a personal risk to the participant.
* Use of medications that may affect the study results.
* Unstable body weight for 3 months prior to the start of the study (> 4 kg loss or gain in weight).
* Active tobacco abuse or illicit drug use, or history of treatment for alcohol abuse.
* On a special diet or prescribed for other reasons (e.g., celiac disease).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Performance | 60min
  Performance measured through the countermovement jump
Performance | 60min
  Deep squat test at 70% of repetition maximum

SECONDARY OUTCOMES:
Heart rate | 60min
  Heart rate will be measured with the Polar H10 heart rate monitor
Subjective fatigue throughe the RPE scale | 60min
  Rate of perceived exertion scale
Recovery | 60min
  Perceived Recovery Status Scale (RPS)
Delayed-onset muscle soreness (DOMS) | 60min
  Delayed-onset muscle soreness (DOMS) scale (0-10 arbitrary units)
Capillar lactate levels | 60min
  Capillar lactate levels
Performance: Weight used in the crosstraining session | 60min
  Weight used in the crosstraining session
Performance: Time performed in the crosstraining session | 60min
  Time performed in the crosstraining session

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de la Laguna, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Undecided